CLINICAL TRIAL: NCT06022146
Title: TB YOUTH - TB sYstemic Management Using One-month, Ultra-short TPT Regimen for scHool Contacts
Acronym: TB-YOUTH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB-YOUTH
Record Dates: First submitted 2023-03-23; First posted 2023-09-01 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tuberculosis; Latent Tuberculosis
Keywords: latent tuberculosis; TPT; active screening
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Isoniazid; rifapentine; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1H3P3 regimen of isoniazid and rifapentine 3 times a week for one month (Experimental): 12-dose ultra-short TPT 1H3P3 regimen of isoniazid and rifapentine 3 times a week for one month
  Interventions: Drug: isoniazid and rifapentine
- 3HR regimen of isoniazid and rifampicin once daily for three months (Active Comparator): 3HR regimen of isoniazid and rifampicin once daily for three months
  Interventions: Drug: Rifampin and Isoniazid

INTERVENTIONS:
Drug: isoniazid and rifapentine — 12-dose ultra-short TPT 1H3P3 regimen of isoniazid and rifapentine 3 times a week for 4 weeks
  Other Names: 1H3P3
  Arms: 1H3P3 regimen of isoniazid and rifapentine 3 times a week for one month
Drug: Rifampin and Isoniazid — 3HR regimen of isoniazid and rifampicin once daily for three months
  Other Names: 3HR
  Arms: 3HR regimen of isoniazid and rifampicin once daily for three months

SUMMARY:
This is a prospective, multi-center, open-label, cluster randomized controlled clinical trial conducted in school settings to estimate the non-inferiority effect of 1H3P3 compared with 3HR.

DETAILED DESCRIPTION:
Background： Adolescents are susceptible to tuberculosis. Almost 1.1 million children (aged below 15 years) and another half a million older adolescents (15-19 years) become ill with TB every year. Approximately 5%-10% people infected with TB develop to active disease, which suggest that a great proportion of adolescents remain undiagnosed and unprotected. Undiagnosed cases and school-based transmission contribute to the burden of TB among adolescents. Closing the gap in targeted interventions for TB prevention in schools is essential to break the cycle of transmission and ensure the well-being of school-aged adolescents. However, TB preventive treatment targeted on adolescents are still lacking.

Method： This is a prospective, multicenter, open-label, non-inferiority, cluster randomized controlled clinical trial within the national tuberculosis control program of GuiZhou,China. Close contacts of school tuberculosis index cases are actively screened with QFT(QuantiFERON-TB Gold Plus), chest X-ray, pooled GeneXpert MTB/RIF test of sputum and symptoms. After ruling out active tuberculosis, LTBI students are enrolled to attend a non-inferiority, cluster randomized controlled clinical trial. The students will be given either 3HR or 1H3P3 regimen and followed for two years. Our primary endpoint is culture or GeneXpert MTB/RIF confirmed TB or clinically highly suggested TB. Assume ICC (interclass correlation coefficient) to be 0.05, and the the lost to follow-up rate is 10%, the study will need 1760 subjects per arm to provide 80% power to detect a 20% non-inferiority margin of primary endpoint between the two arms.

Discussion:

The effectiveness of contact investigation among adolescent students as a tool for improved tuberculosis control has not been established. The integration of ultra-short treatment regimens with active screening holds the potential to provide a comprehensive and effective strategy for tuberculosis prevention and control in school environments, which may help reform the national tuberculosis policy regarding adolescent TB.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥13 years and body weight ≥ 30 kg;
2. School-registered individuals including:

   * Currently attending junior / senior high school or university students;
   * School staff members;
3. Close contacts of active pulmonary TB index cases (confirmed or clinically diagnosed) within the school, defined by meeting both of the following:

   * Teachers/students sharing the same classroom or dormitory with the index case;
   * Exposure history: Prolonged sharing of enclosed space (>4 hours total within 1 week) with the index case;
4. Confirmed LTBI status through screening;
5. Voluntary participation with signed informed consent form (for adults ≥18 years);
6. Parental / guardian consent and co-signed informed consent form (for minors aged 13-17 years).

Exclusion Criteria:

1. Current active TB disease (clinically or bacteriologically confirmed);
2. Documented isoniazid/rifampicin resistance in the corresponding M. tuberculosis strain from the index case;
3. Self-reported use of rifamycins (e.g., rifampicin, rifapentine) or isoniazid for >14 consecutive days within the past 2 years;
4. Prior completion of full-course of treatment for ATB or LTBI;
5. Hypersensitivity or intolerance to rifamycins (rifapentine / rifampicin) or isoniazid;
6. HIV positive serostatus or AIDS patients;
7. History of viral hepatitis (e.g., chronic hepatitis B, chronic hepatitis C) or liver cirrhosis;
8. Liver dysfunction (TBil>2.5mg/dL [43umol/L] or ALT / AST>2ULN) or renal dysfunction.
9. Current receiving immunosuppressive therapy or biological agents.
10. Hematologic disorders with either PLT<50×109/L or WBC<3.0×109/L.
11. Other conditions deemed unsuitable for TPT by investigators.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3520 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with culture or GeneXpert MTB/RIF confirmed TB or clinically highly suggested TB | up to 24 months after randomization
  The primary aim is to estimate the effectiveness non-inferiority of 1H3P3 to 3HR.

SECONDARY OUTCOMES:
Number of participants permanently withdrawal from medication for any reason. | up to 24 months after randomization
  subjects may withdrawal from medication after serious adverse effect
Number of participants complete the treatment. | up to 24 months after randomization
  to compare the completion rates of the two regimens
All-cause mortality. | up to 24 months after randomization
  subjects may withdrawal from this study because of death
Number of participants with drug resistance result. | up to 24 months after randomization
  to study drug resistance condition of school TB endemic

OTHER OUTCOMES:
Patient Report Outcome | from baseline to 1 month after treatment
  health state utility and EuroQol visual analogue scale values measured by ED-5D-3L questionnaire

CONTACTS AND LOCATIONS:
Locations (46):
- China (46):
  - People's Hospital of Hezhang, Bijie, Guizhou
  - People's Hospital of Qianxi, Bijie, Guizhou
  - People's Hospital of Weining, Bijie, Guizhou
  - People's Hospital of Zhijin, Bijie, Guizhou
  - People's Hospital of Daozhen Klau and Hmong autonomous county, Daozhen Klau and Hmong Autonomous County in Zun'yi, Guizhou
  - Liuzhi Special District, Liupanshui, Guizhou
  - People's Hospital of Panzhou, Liupanshui, Guizhou
  - People's Hospital of Shuicheng District, Liupanshui City, Liupanshui, Guizhou
  - Second People's Hospital of Liupanshui City, Liupanshui, Guizhou
  - Third People's Hospital of Liupanshui, Liupanshui, Guizhou
  - People's Hospital of Cengong, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - People's Hospital of Congjiang, Qiandongnan Miao and Dong Autonomous Prefecture, Guizhou
  - First People's Hospital of Kaili, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Danzhai, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Huangping, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Jianhe, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Jinping, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Liping, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Rongjiang, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Sansui, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Shibing, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Tianzhu, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - People's Hospital of Zhenyuan, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - Poeple's Hospital of Leishan, Qiandongnan Miao and Dong Autonomous Region, Guizhou
  - Guizhou Aerospace Hospital, Zunyi, Guizhou
  - People's Hospital of Bozhou District, Zunyi, Guizhou
  - People's Hospital of Chishui, Zunyi, Guizhou
  - People's Hospital of Fenggang, Zunyi, Guizhou
  - People's Hospital of Honghuagang District, Zunyi, Guizhou
  - People's Hospital of Meitan, Zunyi, Guizhou
  - People's Hospital of Renhuai, Zunyi, Guizhou
  - People's Hospital of Suiyang, Zunyi, Guizhou
  - People's Hospital of Tongzi, Zunyi, Guizhou
  - People's Hospital of Wuchuan Klau and Hmong autonomous county, Zunyi, Guizhou
  - People's Hospital of Xishui, Zunyi, Guizhou
  - People's Hospital of Yuqing, Zunyi, Guizhou
  - People's Hospital of Zhengan, Zunyi, Guizhou
  - Zunyi Infectious Disease Hospital, Zunyi, Guizhou
  - Dalian Public Health Clinical Center, Dalian, Liaoning
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - 3rd People's Hospital of Bijie, Bijie
  - People's Hospital of Dafang Town, Bijie
  - People's Hospital of Nayong, Bijie
  - Chinese Medicine Hospital of Qingzhen, Guiyang
  - People's Hospital of Majiang, Qiandongnan Miao and Dong Autonomous Region
  - People's Hospital of Taijiang, Qiandongnan Miao and Dong Autonomous Region

IPD SHARING:
Plan to Share IPD: No
This research targets adolescent students in school. We decide not to share IPD from the ethical perspective.

REFERENCES:
- [Derived] Ruan QL, Yang QL, Ma CL, Lin MY, Huang XT, Mao YP, Gao JM, Li JJ, Zhang XN, You ZX, Zheng QQ, Ren YF, Liu XF, Shao LY, Zhang WH. Efficacy and safety of a novel short course rifapentine and isoniazid regimen for the preventive treatment of tuberculosis in Chinese silicosis patients: a pilot study (SCRIPT-TB). Emerg Microbes Infect. 2025 Dec;14(1):2502010. doi: 10.1080/22221751.2025.2502010. Epub 2025 May 16. PMID 40326358